CLINICAL TRIAL: NCT02482805
Title: Effect of Hormones on Response to Exposure Therapy for Social Anxiety Disorder
Brief Title: Hormones and Social Anxiety Disorder Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SAD - Hormones
Record Dates: First submitted 2015-06-17; First posted 2015-06-26 (Estimated); Results first posted 2017-10-16 (Actual); Last update posted 2017-11-24 (Actual); Status verified 2017-10

CONDITIONS: Social Anxiety Disorder
MeSH Terms: conditions — Phobia, Social | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Power Posing (Experimental): Individuals hold two, 1-minute postures associated with dominance and high power prior to exposure therapy.
  Interventions: Behavioral: Cognitive Behavioral Therapy
- Submissive Posing (Experimental): Individuals hold two, 1-minute postures associated with submissiveness and low power prior to exposure therapy.
  Interventions: Behavioral: Cognitive Behavioral Therapy
- Rest (Experimental): Individuals rest (no postures) for 2 minutes prior to exposure therapy.
  Interventions: Behavioral: Cognitive Behavioral Therapy

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy — Exposure therapy for social anxiety disorder

SUMMARY:
The purpose of this study is to determine whether power posing (i.e., holding poses associated with dominance and power), compared to submissive posing or rest, prior to exposure therapy for social anxiety disorder: 1) leads to a temporary increase in testosterone levels and/or 2) facilitates exposure therapy outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients between the ages of 18 to 70 years of age with a primary psychiatric diagnosis (designated by the patient as the most important source of current distress) of social anxiety disorder as defined by DSM-5 criteria, with fear of public speaking endorsed as a primary concern.
* Willingness and ability to participate in the informed consent process and comply with the requirements of the study protocol.

Exclusion Criteria:

* Current use of testosterone enhancing products (i.e., gels, creams, or injections)
* A lifetime history of bipolar disorder, schizophrenia, psychosis, or delusional disorders; organic brain syndrome, mental retardation or other cognitive dysfunction that could interfere with capacity to engage in therapy; a history of substance or alcohol abuse or dependence (other than nicotine) in the last 6 months.
* Entry of patients with other mood or anxiety disorders will be permitted in order to increase accrual of a clinically relevant sample; however in cases where SAD is not judged to be the predominant disorder, participants will not be eligible.
* Patients with significant suicidal ideation or who have enacted suicidal behaviors within 6 months prior to intake will be excluded from study participation and referred for appropriate clinical intervention.
* Patients using psychotropic medication (e.g., antidepressants, anxiolytics, beta blockers) must be on a stable dose for three weeks prior to initiation of randomized treatment.
* Significant personality dysfunction likely to interfere with study participation.
* Patients with a current or past history of seizures.
* Any concurrent psychotherapy initiated within 3 months of baseline, or ongoing psychotherapy of any duration directed specifically toward treatment of the SAD is excluded. Prohibited psychotherapy includes CBT or psychodynamic therapy focusing on exploring specific, dynamic causes of the phobic symptomatology and providing management skills. General supportive therapy initiated > 3 months prior is acceptable.
* Prior non-response to adequately delivered exposure (i.e., as defined by the patient's report of receiving specific and regular exposure assignments as part of a previous treatment).
* Patients with a history of head trauma causing loss of consciousness, seizure or ongoing cognitive impairment.
* Subjects with back pain issues or medical conditions that would make it difficult to hold posture manipulations.
* Insufficient command of the English language.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2015-07; Primary Completion 2016-12 (Actual); Study Completion 2017-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Texas at Austin, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Power Posing | Submissive Posing | Rest
Started | 26 | 27 | 20
Completed | 22 | 23 | 20
Not Completed | 4 | 4 | 0
Not completed — Lost to Follow-up | 4 | 4 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Power Posing | Submissive Posing | Rest | Total
Number analyzed (Participants) | 26 | 27 | 20 | 73
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.88 (6.99) | 25.26 (8.99) | 24.60 (5.83) | 25.66 (7.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 18 | 16 | 52
  Male | 8 | 9 | 4 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 9 | 3 | 17
  Not Hispanic or Latino | 20 | 17 | 16 | 53
  Unknown or Not Reported | 1 | 1 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 6 | 5 | 3 | 14
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 2 | 3 | 7
  White | 14 | 14 | 11 | 39
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 4 | 6 | 3 | 13
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 26 | 27 | 20 | 73
LSAS-performance [Mean (Standard Deviation); unit: units on a scale] — The Liebowitz Social Anxiety Scale (LSAS) - Performance Subscale is a subscale of a common measure of social anxiety symptom severity. This subscale consists of only 13 (of the total 24) items related to performance situations. Participants rate both their fear (0 to 3) and avoidance (0 to 3) of these 13 situations, where higher scores indicate worse social anxiety severity. The minimum possible score on this subscale is 0 and the maximum possible score is 78.
  units on a scale | 37.96 (14.39) | 36.19 (10.92) | 37.85 (10.16) | 37.27 (11.96)
Peak SUDS during exposure [Mean (Standard Deviation); unit: units on a scale] — Peak Subjective Units of Distress Scale (SUDS) is the maximum amount of fear experienced rated on a 0 to 100 point scale, where 0 indicates no anxiety and 100 indicates the maximum level of anxiety.
  units on a scale | 76.31 (14.86) | 77.74 (15.03) | 77.50 (11.20) | 77.16 (13.85)

OUTCOME MEASURES:

1. Primary Outcome: LSAS-performance Subscale
Description: Liebowitz Social Anxiety Scale (LSAS)-Performance Subscale at pre- and 1-week post-treatment.
  The Liebowitz Social Anxiety Scale (LSAS) - Performance Subscale is a subscale of a common measure of social anxiety symptom severity. This subscale consists of only 13 (of the total 24) items related to performance situations. Participants rate both their fear (0 to 3) and avoidance (0 to 3) of these 13 situations, where higher scores indicate worse social anxiety severity. The minimum possible score on this subscale is 0 and the maximum possible score is 78.
Time Frame: Scores at 1 week post-treatment
Population: 4 individuals did not complete LSAS at post-treatment; accordingly the analyses were conducted with only 69 individuals (versus the total sample size of 73) who had complete data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Power Posing | Submissive Posing | Rest
Number analyzed (Participants) | 23 | 26 | 20
units on a scale | 34.04 (14.76) | 32.54 (8.74) | 32.05 (13.70)

2. Primary Outcome: Subjective Units of Distress Scale (SUDs)
Description: Peak (max) SUDS ratings (0 to 100 scale) during treatment exposure and 1 week post-treatment exposure.
  Peak Subjective Units of Distress Scale (SUDS) is the maximum amount of fear experienced rated on a 0 to 100 point scale, where 0 indicates no anxiety and 100 indicates the maximum level of anxiety.
Time Frame: Scores at 1 week post-treatment
Population: 8 individuals did not complete the post-treatment exposure; accordingly the analyses were conducted with only 66 individuals (versus the total sample size of 73) who had complete data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Power Posing | Submissive Posing | Rest
Number analyzed (Participants) | 23 | 23 | 20
units on a scale | 59.26 (14.43) | 59.17 (23.85) | 48.75 (19.79)

3. Primary Outcome: Salivary Testosterone Levels
Description: Saliva sample taken before posture manipulation and 20 minutes after. Outcome is the change from pre- to post-manipulation in testosterone levels.
Time Frame: Baseline and 20 minutes after posture manipulation
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Power Posing | Submissive Posing | Rest
Number analyzed (Participants) | 26 | 27 | 20
pg/mL | -2.31 (10.82) | -0.88 (33.31) | -1.47 (54.56)

ADVERSE EVENTS:
Arm/Group | Power Posing | Submissive Posing | Rest
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/27 | 0/20
Other Adverse Events (participants affected / at risk) | 0/26 | 0/27 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No